CLINICAL TRIAL: NCT05694156
Title: Musical Attention Control and Executive Function Training for Adults With MDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBCT-01
Record Dates: First submitted 2022-12-27; First posted 2023-01-23 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder; Cognitive Dysfunction; Suicide
Keywords: music-based intervention; cognition; depression
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction; Suicide; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Music-based cognitive training (Experimental): Music-based cognitive training sessions are derived from two Neurologic Music Therapy techniques: Musical Attention Control Training (MACT) and Musical Executive Function Training (MEFT). MACT exercises will focus on sustained and selective attention to emphasise flexibility and adaptability of the auditory attention system. MEFT exercises will provide opportunity for decision making, problem solving, reasoning, comprehending, organising, initiating, inhibiting, evaluating, analysing, and creating.
  Interventions: Other: Music-based cognitive training

INTERVENTIONS:
Other: Music-based cognitive training — 8-week music-based cognitive training

SUMMARY:
The investigators have developed music-based cognitive training sessions derived from Neurologic Music Therapy (NMT) techniques. The music-based cognitive training sessions will address areas of attention and executive function, which appear to progress over time and worsen as an individual experiences more episodes of depression. The aim of this pilot is to test 8-weeks of music-based cognitive training to improve cognitive function among adults with major depressive disorder.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a lifelong condition and is the leading cause of disability in the world. MDD is a multifaceted mood disorder and due to its complex nature, this mental health diagnosis affects emotional, behavioural, and cognitive processing. Cognitive dysfunction appears to progress over time and worsens as the individual experiences more episodes of depression. Because of this, it is critical to continue to investigate and formulate effective treatment that can target and improve not only depressive symptoms, but also address overall cognitive function. Thus, the investigators propose implementing music-based cognitive training derived from Neurologic Music Therapy (NMT) techniques to address cognitive dysfunction experienced by adults diagnosed with MDD. Music-based interventions, specifically from the NMT approach have been shown to physically change the human brain when working on cognition in areas of attention and executive function, however little is known of these applications with adults with MDD. The aim of this pilot is to test 8-weeks of music-based cognitive training to improve cognitive function among adults with MDD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MDD meeting the Diagnostic and Statistical Manual Diploma in Social Medicine (DSM-V) criteria
* Experiencing suicidal ideation in the past week (Beck Scale for Suicide Ideation >10)
* Have received more than 12 sessions of psychotherapy
* Stable medication use > 4 weeks
* Ability to undergo music-based cognitive training sessions in English
* Capable of giving informed consent

Exclusion Criteria:

* The presence of cognitive impairment that would limit consent or understanding of neurologic music therapy
* The presence of active psychosis
* The presence of mood and suicidal symptom severity requiring immediate treatment
* Hearing impairment
* Participation in music therapy 6 months prior to study
* Private music lessons for a period of 1 year prior to study
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Change in inhibition using the Go/No Go Task | From baseline to 8-weeks
  This cognitive task measures response time, accuracy, commission errors, omission errors, and reaction time variability.
Change in working memory capacity using the Digit Span Forward and Backward Test | From baseline to 8-weeks
  This cognitive task measures span length, correct recall, error rate, and reaction time.
Change in cognitive flexibility and executive control using the Shifting Attention test | From baseline to 8-weeks
  This cognitive task measures the ability to shift attention between different stimuli, assessing the speed and accuracy with which the individual can shift their attention and switch between different rules.
Change in visual attention and task switching using the Trail Making A and B test | From baseline to 8-weeks
  This cognitive task measures the time to complete the task and errors made.
  In Trail Making Test A, a longer completion time and higher number of errors can indicate difficulties with processing speed and attention.
  In Trail Making Test B, a longer completion time and a higher number of errors on Trail Making Test B, compared to Trail Making Test A, can indicate difficulties with cognitive flexibility, mental shifting, and attention.
Change in selective attention using the Stroop Test | From baseline to 8-weeks
  This cognitive task measures the time to complete the task and errors made. A longer completion time and a higher number of errors can indicate difficulty with selective attention and mental flexibility.

SECONDARY OUTCOMES:
Change in suicidal ideation using the Beck Scale for Suicide Ideation (BSSI) | From baseline to 8-weeks
  A 21-item self-report scale that quantifies suicidal ideation. The BSSI is a Likert-style questionnaire, where each item is rated on a scale from 0 to 3, with higher scores indicating a greater severity of suicidal thoughts and behaviours. The minimum possible score on the BSSI is 0, which would indicate the absence of suicidal ideation. The maximum possible score is 63, which would indicate a high level of severity of suicidal thoughts and behaviours.
Changes in affect using the Positive and negative affect schedule - short form (PNAS-SF) | From baseline to 8-weeks
  A 10-item scale to assess the experience of positive and negative emotions/feelings. Each item is rated on a 5-point Likert scale, ranging from 1 (very slightly or not at all) to 5 (extremely).
  The minimum possible score on the PNAS-SF for positive affect is 10, which would indicate the absence of positive affect. The maximum possible score is 50, which would indicate a high level of positive affect.
  The minimum possible score on the PNAS-SF for negative affect is 10, which would indicate the absence of negative affect. The maximum possible score is 50, which would indicate a high level of negative affect.
Changes in depression symptoms using the Quick Inventory of Depressive Symptomatology - self-report (QIDS-SR). | From baseline to 8-weeks
  A 16-item validated depression scale. Each item is rated on a 4-point Likert scale, ranging from 0 (not at all) to 3 (severe).
  The minimum possible score on the QID-SR is 0, which would indicate the absence of depression. The maximum possible score is 48, which would indicate a high level of depression severity.
Changes in quality of life using the Quality of Life Scale (QOLS) | From baseline to 8-weeks
  A validated 16-item scale to assess quality of life. Each item is rated on a 7-point Likert scale , ranging from 1 (terrible) to 7 (delighted).
  The minimum possible score on the QOLS is 16, which would indicate poor quality of life. The maximum possible score is 112, which would indicate excellent quality of life.
Feasibility and acceptability of music-based cognitive training | From baseline to 8-weeks
  Feasibility and Acceptability survey and interview created in-house with questions designed to collect quantitative and qualitative feedback from participants with respect to the feasibility and acceptability of the music-based cognitive training intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sakina Rizvi, PhD,MACP,RP, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schoonees R, de Klerk JN, Murphy GP. The effect of prolactin on organ weights and zinc-65 uptake in male baboons. J Surg Oncol. 1970;2(2):103-6. doi: 10.1002/jso.2930020204. No abstract available. PMID 4999943
- [Background] Pan Z, Park C, Brietzke E, Zuckerman H, Rong C, Mansur RB, Fus D, Subramaniapillai M, Lee Y, McIntyre RS. Cognitive impairment in major depressive disorder. CNS Spectr. 2019 Feb;24(1):22-29. doi: 10.1017/S1092852918001207. Epub 2018 Nov 23. PMID 30468135
- [Background] McIntyre RS, Soczynska JZ, Woldeyohannes HO, Alsuwaidan MT, Cha DS, Carvalho AF, Jerrell JM, Dale RM, Gallaugher LA, Muzina DJ, Kennedy SH. The impact of cognitive impairment on perceived workforce performance: results from the International Mood Disorders Collaborative Project. Compr Psychiatry. 2015 Jan;56:279-82. doi: 10.1016/j.comppsych.2014.08.051. Epub 2014 Aug 23. PMID 25439523
- [Background] Thaut MH, Gardiner JC, Holmberg D, Horwitz J, Kent L, Andrews G, Donelan B, McIntosh GR. Neurologic music therapy improves executive function and emotional adjustment in traumatic brain injury rehabilitation. Ann N Y Acad Sci. 2009 Jul;1169:406-16. doi: 10.1111/j.1749-6632.2009.04585.x. PMID 19673815
- [Background] Hsu WC, Lai HL. Effects of music on major depression in psychiatric inpatients. Arch Psychiatr Nurs. 2004 Oct;18(5):193-9. doi: 10.1016/j.apnu.2004.07.007. PMID 15529285
- [Background] Keilp JG, Gorlyn M, Russell M, Oquendo MA, Burke AK, Harkavy-Friedman J, Mann JJ. Neuropsychological function and suicidal behavior: attention control, memory and executive dysfunction in suicide attempt. Psychol Med. 2013 Mar;43(3):539-51. doi: 10.1017/S0033291712001419. Epub 2012 Jul 10. PMID 22781400
- [Background] Lam RW, Kennedy SH, Mclntyre RS, Khullar A. Cognitive dysfunction in major depressive disorder: effects on psychosocial functioning and implications for treatment. Can J Psychiatry. 2014 Dec;59(12):649-54. doi: 10.1177/070674371405901206. No abstract available. PMID 25702365
- [Background] Strait DL, Kraus N. Can you hear me now? Musical training shapes functional brain networks for selective auditory attention and hearing speech in noise. Front Psychol. 2011 Jun 13;2:113. doi: 10.3389/fpsyg.2011.00113. eCollection 2011. PMID 21716636
- [Background] Strait DL, Slater J, O'Connell S, Kraus N. Music training relates to the development of neural mechanisms of selective auditory attention. Dev Cogn Neurosci. 2015 Apr;12:94-104. doi: 10.1016/j.dcn.2015.01.001. Epub 2015 Jan 13. PMID 25660985
- [Background] Thaut MH, McIntosh GC, Hoemberg V. Neurobiological foundations of neurologic music therapy: rhythmic entrainment and the motor system. Front Psychol. 2015 Feb 18;5:1185. doi: 10.3389/fpsyg.2014.01185. eCollection 2014. PMID 25774137
- [Background] Zatorre RJ. Musical pleasure and reward: mechanisms and dysfunction. Ann N Y Acad Sci. 2015 Mar;1337:202-11. doi: 10.1111/nyas.12677. PMID 25773636
- [Background] Culpepper L, Lam RW, McIntyre RS. Cognitive Impairment in Patients With Depression: Awareness, Assessment, and Management. J Clin Psychiatry. 2017 Nov/Dec;78(9):1383-1394. doi: 10.4088/JCP.tk16043ah5c. PMID 29345866
- [Background] Knight MJ, Baune BT. Executive Subdomains Are Differentially Associated With Psychosocial Outcomes in Major Depressive Disorder. Front Psychiatry. 2018 Jul 10;9:309. doi: 10.3389/fpsyt.2018.00309. eCollection 2018. PMID 30042703